CLINICAL TRIAL: NCT01227213
Title: The Vascular and Metabolic Effects of Sunitinib in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, G. Rongen, Prof. dr. Rongen, Radboud University Medical Center
Other Study IDs: SUMAVA
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension; Renal Function; Insulin Sensitivity; Renal Cell Carcinoma
MeSH Terms: conditions — Hypertension; Insulin Resistance; Carcinoma, Renal Cell

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: The introduction of angiogenesis inhibitors, like sunitinib and bevacizumab, has improved the outcome of patients with several types of cancer remarkably. However, their application is hampered by side effects, such as development of hypertension with consequences for renal and cardiac function. Moreover patients treated with angiogenesis inhibitors may suffer from weight loss, and insulin sensitivity during treatment appears to change. The treatment with angiogenesis inhibitors, will improve life expectancy of patients with various cancer diagnoses and therefore the clinical relevance of both short term and long lasting adverse events will translate into reduced quality of life. In addition, premature withdrawal of angiogenesis inhibitors due to side effects may result in lower response, shorter duration of response and possibly a shorter survival. Therefore, adequate treatment of above mentioned side effects in patients treated with angiogenesis inhibitors is of relevance for the response rate, the duration of progression free survival and overall survival and for quality of life.

Mechanistic insight in the pathogenesis of these side effects will help optimizing treatment.

Objective: The primary objective of the study is to investigate the effect of sunitinib on endothelial function, insulin sensitivity, renal function and renal blood flow.

Study design: Single-centre non randomized observational study Study population: 30 Patients (>18 years old) starting with sunitinib as treatment for metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form
* Age 18 years or older
* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* mRCC patients in which the treatment of choice is sunitinib

Exclusion Criteria:

* Use of corticosteroids
* Any evidence of severe or uncontrolled diseases other than renal cell carcinoma eg, unstable or uncompensated respiratory, cardiac, hepatic or renal disease.
* Known risk of the patient transmitting HIV, hepatitis B or C via infected blood
* Patients being treated with oral anticoagulants if to be included in group A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with metastatic renal cell carcinoma starting treatment with sunitinib
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 2 weeks
  Group A:
  Vasomotor response to intra-arterially administered doses of acetylcholine and nitroprusside before and after start sunitinib
Insulin sensitivity | 2 weeks
  Group B:
  Insulin sensitivity measured by hyperinsulinemic euglycemic clamp before and after start sunitinib
GFR and renal perfusion flow | 2 weeks
  Group C:
  GFR and RPF measured by PAH and inulin clearance before and after start of treatment with sunitinib

SECONDARY OUTCOMES:
Blood pressure | 3 months
Weight | 3 months
Laboratory evaluations | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Thijs AM, van Herpen CM, Verweij V, Pertijs J, van den Broek PH, van der Graaf WT, Rongen GA. Impaired endothelium-dependent vasodilation does not initiate the development of sunitinib-associated hypertension. J Hypertens. 2015 Oct;33(10):2075-82. doi: 10.1097/HJH.0000000000000662. PMID 26203967
- [Result] Thijs AM, Tack CJ, van der Graaf WT, Rongen GA, van Herpen CM. The early effect of sunitinib on insulin clearance in patients with metastatic renal cell carcinoma. Br J Clin Pharmacol. 2016 Apr;81(4):768-72. doi: 10.1111/bcp.12797. Epub 2016 Jan 14. PMID 26447463